CLINICAL TRIAL: NCT01025284
Title: A Phase 2 Study of LY2523355 in Patients With Extensive-Stage Small-Cell Lung Cancer
Brief Title: A Study for Participants With Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12253; I1Y-MC-JFBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — litronesib; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A LY2523355 (Experimental): 8 milligrams per square meter (mg/m²) per dose based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 5, 9 of each 21-day cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: LY2523355
- Part B LY2523355 (Experimental): 5 or 6 mg/m² per dose based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 2, 3 plus granulocyte colony-stimulating factor (G-CSF) support administered subcutaneously beginning on Day 4 of each 21-day cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: LY2523355; Drug: Granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: LY2523355 — Administered intravenously as a 1-hour infusion
Drug: Granulocyte colony-stimulating factor (G-CSF) — Administered subcutaneously
  Arms: Part B LY2523355

SUMMARY:
Part A: This study evaluates an experimental treatment in participants with extensive-disease in small-cell lung cancer.

Part B: This study evaluates an experimental treatment in participants with extensive-disease in small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of extensive-disease small-cell lung cancer
* Have the presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Have received at least 1 prior chemotherapy regimen with agents known to provide clinical benefit for small-cell lung cancer and be, in the opinion of the investigator, an appropriate candidate for experimental therapy
* Have discontinued all previous therapies for cancer, including chemotherapy, biologic therapy, hormone therapy, or radiotherapy. Participants must have recovered from the acute effects of therapy (except alopecia and fatigue) before study enrollment
* Part A: Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group scale
* Part B: Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group scale

Exclusion Criteria:

* Have received treatment within 28 days of the first dose of LY2523355 with a drug that has not received regulatory approval for any indication
* Have a mixed histological diagnosis of small-cell lung cancer and non-small-cell lung cancer
* Have serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in this study
* Part A: Have symptomatic, untreated, or uncontrolled central nervous system (CNS) metastases. Participants with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and corticosteroid use has been discontinued for at least 2 weeks prior to the first dose of study drug. Screening of asymptomatic participants without history of CNS metastases is not required
* Part B: Have symptomatic, untreated, or uncontrolled CNS metastases or a history of CNS metastases. Participants who have received prophylactic radiation are not excluded. Screening of asymptomatic participants without history of CNS metastases is not required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time(UTC/GMT-5hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrington, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scarborough, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a nonrandomized, open-label, 2-part study.
Groups:
- Part A - 8 mg/m²/Day: 8 milligrams per square meter (mg/m²) of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of each 21-day cycle.
- Part B - 5 mg/m²/Day: 5 mg/m² of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 2, and 3 plus granulocyte colony-stimulating factor (G-CSF) support given per local package insert beginning on Day 4 of each 21-day cycle.
- Part B - 6 mg/m²/Day: 6 mg/m² of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 2, and 3 plus G-CSF support given per local package insert beginning on Day 4 of each 21-day cycle.
Period: Overall Study
Arm/Group | Part A - 8 mg/m²/Day | Part B - 5 mg/m²/Day | Part B - 6 mg/m²/Day
Started | 38 | 18 | 8
Received at Least 1 Dose of Study Drug | 38 | 18 | 8
Completed | 38 | 16 | 8
Not Completed | 0 | 2 | 0
Not completed — Investigator Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - 8 mg/m²/Day | Part B - 5 mg/m²/Day | Part B - 6 mg/m²/Day | Total
Number analyzed (Participants) | 38 | 18 | 8 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.88 (6.3) | 63.33 (8.4) | 63.40 (9.1) | 64.26 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 2 | 16
  Male | 27 | 15 | 6 | 48
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 12 | 5 | 4 | 21
  Black or African American | 1 | 0 | 1 | 2
  White | 25 | 13 | 3 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 10 | 4 | 31
  Romania | 9 | 3 | 0 | 12
  South Korea | 12 | 5 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Achieving an Overall Response (Overall Response Rate)
Description: The overall response is complete response (CR) + partial response (PR) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions. The overall response rate is calculated as a total number of participants with CR or PR, then divided by the total number of participants treated, then multiplied by 100.
Time Frame: Date of enrollment to date of measured progressive disease up to 99.6 weeks
Population: All participants who received at least 1 dose of study drug in Part A.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Part A: 8 milligrams per square meter (mg/m²) of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of each 21-day cycle.
Arm/Group | Part A
Number analyzed (Participants) | 38
percentage of participants | 2.6 [0.1 to 11.9]

2. Primary Outcome: Part B: Percentage of Participants Achieving a Best Response (Clinical Benefit Rate)
Description: Clinical benefit rate is complete response (CR) + partial response (PR) + stable disease (SD) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Clinical benefit rate is calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated, then multiplied by 100.
Time Frame: Date of enrollment to date of measured progressive disease up to 18.1 weeks
Population: All participants who received at least 1 dose of study drug in Part B.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Part B: 5 or 6 milligrams per square meter (mg/m²) of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 2, and 3 plus granulocyte colony-stimulating factor (G-CSF) support given per local package insert beginning on Day 4 of each 21-day cycle.
Arm/Group | Part B
Number analyzed (Participants) | 26
percentage of participants | 26.9 [13.4 to 44.7]

3. Secondary Outcome: Part A: Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the time from the date of enrollment (first treatment dose) to the first observation of progression of disease (PD) or death due to any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD is a ≥20% increase in sum of longest diameter of target lesions and/or a new lesion. For participants who had no PD or death or starting new anti-cancer therapy, PFS was censored at their last radiological tumor assessment.
Time Frame: Date of enrollment to date of measured progressive disease or date of death from any cause up to 99.6 weeks
Population: All participants who received at least 1 dose of study drug in Part A. The numbers of participants censored are 4.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Part A
Number analyzed (Participants) | 38
weeks | 5.3 [5.1 to 5.7]

4. Secondary Outcome: Part B: Progression-Free Survival
Description: as for outcome 3
Time Frame: Date of enrollment to date of measured progressive disease or date of death from any cause up to 18.1 weeks
Population: All participants who received at least 1 dose of study drug in Part B. The numbers of participants censored are 4.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Part B
Number analyzed (Participants) | 26
weeks | 6.1 [5.6 to 7.4]

5. Secondary Outcome: Part A: Percentage of Participants Achieving a Best Response (Clinical Benefit Rate)
Description: as for outcome 2
Time Frame: Date of enrollment to date of measured progressive disease 99.6 weeks
Population: All participants who received at least 1 dose of study drug in Part A.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A
Number analyzed (Participants) | 38
percentage of participants | 23.7 [12.9 to 37.7]

6. Secondary Outcome: Part B: Percentage of Participants Achieving an Overall Response (Overall Response Rate)
Description: The overall response is complete response (CR) + partial response (PR) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions. The overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants treated, then multiplied by 100.
Time Frame: Date of enrollment to date of measured progressive disease up to 18.1 weeks
Population: All participants who received at least 1 dose of study drug in Part B.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part B
Number analyzed (Participants) | 26
percentage of participants | 0 [NA to NA] — No participants had CR or PR, therefore 90% Confidence Interval was not calculable.

7. Secondary Outcome: Part A: Pharmacokinetics - Maximum Observed Plasma Concentration (Cmax) of LY2523355 and Its Metabolite (LSN2546307)
Time Frame: Days 1,5 and 9 of Cycle 1 (21-day cycle)
Population: All participants who received 1 dose of study drug on Days 1, 5, and 9 of Cycle 1 and had Cmax samples collected on Days 1, 5, and 9 of Cycle 1 in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Part A
Number analyzed (Participants) | 37
nanograms/milliliter (ng/mL)
  LY2523355 Day 1 | 146 (69.5)
  LY2523355 Day 5: number analyzed (Participants) | 34
  LY2523355 Day 5 | 157 (91.4)
  LY2523355 Day 9: number analyzed (Participants) | 14
  LY2523355 Day 9 | 100 (420)
  Metabolite Day 1 | 7.17 (55.4)
  Metabolite Day 5: number analyzed (Participants) | 34
  Metabolite Day 5 | 6.29 (50.8)
  Metabolite Day 9: number analyzed (Participants) | 14
  Metabolite Day 9 | 6.11 (129)

8. Secondary Outcome: Part B: Pharmacokinetics - Maximum Observed Plasma Concentration (Cmax) of LY2523355
Time Frame: Day 3 of Cycle 1 (21-day cycle)
Population: All participants who received 1 dose of study drug on Days 1, 2, and 3 of Cycle 1 and had Cmax samples collected on Day 3 of Cycle 1 in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Part B - 5 mg/m²/Day: 5 milligrams per square meter (mg/m²) of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 2, and 3 plus granulocyte colony-stimulating factor (G-CSF) support given per local package insert beginning on Day 4 of each 21-day cycle.
Arm/Group | Part B - 5 mg/m²/Day | Part B - 6 mg/m²/Day
Number analyzed (Participants) | 17 | 6
nanograms/milliliter (ng/mL) | 128 (82) | 258 (32)

9. Secondary Outcome: Part A: Pharmacokinetics - Area Under the Plasma Concentration Versus Time Curve of LY2523355 From Time Zero to Infinity [AUC(0-∞)]
Description: Due to the very limited pharmacokinetic sampling employed in Part A of the study, the AUC(0-∞) of LY2523355 could not be accurately calculated.
Time Frame: Days 1,5 and 9 of Cycle 1 (21-day cycle)
Population: No participants were analyzed due to the very limited pharmacokinetic sampling employed in Part A that did not allow accurate calculation of the AUC(0-∞) on Days 1, 5, and 9 of Cycle 1.
Arm/Group | Part A
Number analyzed (Participants) | 0

10. Secondary Outcome: Part B: Pharmacokinetics - Area Under the Plasma Concentration Versus Time Curve of LY2523355 From Time Zero to Infinity [AUC(0-∞)]
Time Frame: Day 3 of Cycle 1 (21-day cycle)
Population: All participants who received 1 dose of study drug on Days 1, 2, and 3 of Cycle 1 and had pharmacokinetic samples collected on Day 3 of Cycle 1 in Part B that enabled calculation of the AUC(0-∞).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- Part B - 6 mg/m²/Day: 6 mg/m² of LY2523355 per day based on participant's body surface area, administered intravenously as a 1-hour infusion on Days 1, 2, and 3 plus granulocyte colony-stimulating factor (G-CSF) support given per local package insert beginning on Day 4 of each 21-day cycle.
Arm/Group | Part B - 5 mg/m²/Day | Part B - 6 mg/m²/Day
Number analyzed (Participants) | 17 | 6
nanograms*hour/milliliter (ng*h/mL) | 639 (41) | 1220 (38)

11. Secondary Outcome: Total Lung Cancer Symptom Scale (LCSS) and Average Symptom Burden Index (ASBI)
Description: LCSS is a 9-item questionnaire. Six questions are symptom-specific measures for lung cancer (appetite, fatigue, cough, dyspnea, hemoptysis and pain), and 3 summation items describe total symptomatic distress, activity status, and overall quality of life. Participant responses were measured using visual analogue scales (VAS) with 100-milliliter (mm) lines. The LCSS total score was defined as the mean of the 9 items of the scale, with scores range from 0 (for best outcome) to 100 (for worst outcome). ASBI was calculated as the mean of six symptom-specific questions from the LCSS, with scores range from 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Baseline and follow-up up to 104 weeks after the first dose of study drug
Population: All participants who received at least 1 dose of study drug and had total LCSS and ASBI scores at baseline and follow-up in Part B.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B
Number analyzed (Participants) | 24
units on a scale
  Total LCSS at Baseline | 28.24 (15.2)
  Total LCSS at Follow-up: number analyzed (Participants) | 16
  Total LCSS at Follow-up | 42.61 (14.5)
  ASBI at Baseline | 26.76 (14.1)
  ASBI at Follow-up: number analyzed (Participants) | 16
  ASBI at Follow-up | 36.41 (11.1)

ADVERSE EVENTS:
Arm/Group | Part A - 8 mg/m²/Day | Part B - 5 mg/m²/Day | Part B - 6 mg/m²/Day
Serious Adverse Events (participants affected / at risk) | 8/38 | 8/18 | 8/8
Other Adverse Events (participants affected / at risk) | 35/38 | 18/18 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 8 mg/m²/Day (N=38) | Part B - 5 mg/m²/Day (N=18) | Part B - 6 mg/m²/Day (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 4 (4)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 2 (3) — Event resulted in a death in Part A
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Event resulted in a death in Part A
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 8 mg/m²/Day (N=38) | Part B - 5 mg/m²/Day (N=18) | Part B - 6 mg/m²/Day (N=8)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 3 (3) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 29 (74) | 11 (17) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (6) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 2 (2) | 3 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (4) | 1 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (2) | 2 (2)
Fatigue (General disorders) | 10 (12) | 7 (9) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (7) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 3 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 3 (3) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days